CLINICAL TRIAL: NCT06734065
Title: Effect of Non-Invasive Lung Fluid Monitoring Using ReDS Technology for Heart Failure Management in Primary Care Settings: A Randomized Controlled Trial
Brief Title: Effect of Non-Invasive Lung Fluid Monitoring for Heart Failure Management in Primary Care
Acronym: LiLAC-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Naoko Perkiö Kato, Associate Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2024-05565-01
Record Dates: First submitted 2024-11-27; First posted 2024-12-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Primary care; Nursing; Monitoring; Self-care; Community
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): Patients in the usual care group will receive usual care.
- ReDS-guided heart failure management group (Experimental)
  Interventions: Behavioral: ReDS-guided heart failure management program

INTERVENTIONS:
Behavioral: ReDS-guided heart failure management program — Remote dielectric sensing (ReDS) system (Sensible Medical Innovations Ltd., Netanya, Israel) is a novel electromagnetic energy-based technology that accurately quantifies changes in lung fluid concentration non-invasively.
  Patients in the intervention group will receive a three-month, ReDS-guided heart failure management program in addition to usual care.
  The program, led by nurses, will integrate algorithms for diuretic use, a structured follow-up schedule, and self-care support tailored to pulmonary fluid levels assessed by ReDS.
  Arms: ReDS-guided heart failure management group

SUMMARY:
Remote dielectric sensing (ReDS) technology offers a non-invasive method for assessing lung congestion. This randomized controlled trial aims to evaluate the effectiveness and processes of the ReDS-guided heart failure management program in primary care settings for patients with heart failure.

DETAILED DESCRIPTION:
Remote dielectric sensing (ReDS) technology offers a non-invasive method for assessing lung congestion. Our newly developed ReDS-guided heart failure management program, led by nurses, incorporates algorithms for a follow-up schedule, diuretic adjustments, and symptom monitoring.

The specific aims of the study are:

1. To examine whether the program decreases the number of urgent healthcare visits for heart failure, unplanned heart failure hospitalisations, and all-cause death in patients with heart failure.
2. To evaluate the intervention processes and explore barriers to and facilitators for the implementation of the program.

This is a multicentre 1:1 randomised controlled clinical trial with a 6-month follow-up. Study participants will be patients with diagnosed with heart failure. The primary outcome will be the total number of urgent healthcare visits for heart failure, unplanned heart failure hospitalisation, and all-cause death at 3 months. Secondary outcomes will include health-related quality of life, self-care behaviour, and healthcare cost. Throughout the randomised controlled trial, a process evaluation will be conducted to assess the fidelity, dose, and reach of the intervention program. Additionally, we will explore both barriers and facilitators for program implementation among study patients and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, there is no upper age limit
* Diagnosed with heart failure regardless of left ventricular ejection fraction
* Having New York Heart Association (NYHA) Class III/IV irrespective of prior hospitalisation for heart failure, or NYHA II with a history of at least one hospitalisation for heart failure within the previous 12 months
* Elevated N-terminal pro-B-type natriuretic peptide (NT-proBNP) within 12 months: (a) ≥450 pg/ml for patients under 50 years; (b) ≥900 pg/ml for patients aged 50-75 years; (c) ≥1800 pg/ml for patients over 75 years.

Exclusion Criteria:

* NYHA I
* Life expectancy <6 months
* Physical characteristics that prevented use of the ReDS (body mass index < 22 or >39, and height less than 155 cm or higher than 195 cm)
* Implantation of a left ventricular assist device or cardiac transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Total number of acute healthcare visits for heart failure, unplanned heart failure hospitalisations, and all-cause death | 3 months

SECONDARY OUTCOMES:
Total number of acute healthcare visits for heart failure | 1 month, 3 months and 6 months
Total number of unplanned hospitalisations for heart failure | 1 month, 3 months and 6 months
Total number of all-cause death | 1 month, 3 months and 6 months
Number of days alive out of hospital | 1 month, 3 months and 6 months
Changes in NT-proBNP/BNP levels | Baseline, 3 months and 6 months
Changes in the remote dielectric sensing (ReDS) values | Baseline, 3 months and 6 months
  The remote dielectric sensing (ReDS) system (Sensible Medical Innovations Ltd., Netanya, Israel) is a novel electromagnetic energy-based technology that accurately quantifies lung fluid content non-invasively. Normal ReDS values range from 20% to 35%. Values above 35% indicate hypervolemia, while values below 20% suggest dehydration.
Changes in the 12-item Kansas City Cardiomyopathy Questionnaire scores | Baseline, 1 month, 3 months and 6 months
  The 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated instrument for quantitatively measuring health status for patients with heart failure. It contains four domains: physical limitation, symptom frequency, quality of life, and social limitations. The KCCQ-12 generates both summary and domain scores ranging from 0 to 100, where 0 represents the worst and 100 the best possible health status.
Changes in the five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) scores | Baseline, 1 month, 3 months and 6 months
  The 5-level EuroQol-5 Dimension version (EQ-5D-5L) assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels, with higher scores indicating better health-related quality of life.
Changes in the heart failrue self-care behaviour scores | Baseline, 1 month, 3 months and 6 months
  The European Heart Failure Self-Care Behaviour Scale (EHFScBS) is a 9-item scale, with higher scores indicating poorer self-care (range: 9-45).

OTHER OUTCOMES:
Healthcare costs | 1 month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Primary care center Centrum Flen, Flen, Sweden

IPD SHARING:
Plan to Share IPD: No